CLINICAL TRIAL: NCT07049107
Title: A Study on the Pharmacokinetic Effects of HRS-8427 Injection on Bupropion and Midazolam in Healthy Subjects
Brief Title: Pharmacokinetics Impact of HRS-8427 on Bupropion and Midazolam in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HRS-8427-105
Record Dates: First submitted 2025-06-24; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Health Volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HRS-8427 (Experimental)
  Interventions: Drug: HRS-8427

INTERVENTIONS:
Drug: HRS-8427 — HRS-8427

SUMMARY:
This study is a single-center, open-label, sequential drug interaction study

The primary objectives are:

To evaluate the pharmacokinetic effects of HRS-8427 injection on the liver drug enzymes CYP2B6 substrate bupropion and CYP3A4 substrate midazolam in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects aged 18 to 45 years old (including 18 and 45 years old, based on the time of signing the informed consent form), both male and female.
2. The weight of female subjects was ≥45 kg, the weight of male subjects was ≥50 kg, and the body mass index (BMI) was within the range of 19.0-26.0 kg/m2
3. The female subjects were not in the pregnancy or lactation period, and the pregnancy examination results before the test were negative; Male or female subjects agreed to take the investigator-approved effective contraceptive measures during the trial as required by the investigator.
4. Before the trial, a thorough understanding of the nature, significance, potential benefits, possible inconveniences and potential risks of the trial was obtained. The participant voluntarily participated in this clinical trial, was able to communicate well with the researcher, comply with the requirements of the entire study, and signed a written informed consent form.

Exclusion Criteria:

1. Those with a history of allergies to food, drugs, etc., especially those known to be allergic to β -lactam antibacterial drugs and midazolam, bupropion, or those with an allergic constitution.
2. Have had or are currently suffering from diseases of the heart, liver, kidneys, endocrine system, digestive tract, immune system, respiratory system, musculoskeletal system and nervous system, etc.
3. Conforming to the contraindications of midazolam use or not suitable for midazolam use .
4. Comply with the contraindications for bupropion use or are not suitable for bupropion use .
5. The 12-lead electrocardiogram was abnormal and was judged by the researcher as unsuitable to participate in this study .
6. Laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), physical examination, vital signs (ears, blood pressure, pulse, respiration), and chest X-ray results, etc., which are judged by clinicians as abnormal and of clinical significance .
7. Those with positive infectious disease tests (human immunodeficiency virus antibody, hepatitis B surface antigen, anti-hepatitis C virus antibody, anti-Treponema pallidum specific antibody).
8. Those who have undergone major surgical operations within the three months prior to screening; Or those who have undergone surgery that may affect the in vivo process or safety evaluation of the studied drug; Or those who plan to undergo surgical operations during the research period.
9. Those who have participated in drug clinical trials as subjects and taken the investigational drug within 3 months prior to screening, or who plan to participate in other clinical trials during this study period .
10. Those who have used any inducers or inhibitors of CYP2B6 and CYP3A enzymes within one month before taking the study drug for the first time.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Cmax | 15 Days
  Bupropion, hydroxybupropion and midazolam, hydroxymidazolam. Observed maximum plasma concentration. Blood samples will be collected.
AUC0-t | 15 Days
  Bupropion, hydroxybupropion and midazolam, hydroxymidazolam. Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. Blood samples will be collected.
AUC0-∞ | 15 Days
  Bupropion, hydroxybupropion and midazolam, hydroxymidazolam. Area under the plasma concentration-time curve from time 0 to infinity. Blood samples will be collected.
Tmax | 15 Days
  Bupropion, hydroxybupropion and midazolam, hydroxymidazolam. Observed time to reach Cmax. Blood samples will be collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided